CLINICAL TRIAL: NCT05553743
Title: The UCSD Human Milk Biorepository
Brief Title: Researchers At UC San Diego Are Learning About the Benefits of Human Milk and How It Influences Infant and Child Health
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christina Chambers, Professor, University of California, San Diego
Other Study IDs: 130658
Record Dates: First submitted 2022-09-19; First posted 2022-09-23 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Breastfeeding; COVID-19 Infection; COVID-19 Vaccine; Remdesivir; Antibiotics
Keywords: Breastfeeding; COVID-19 Infection; COVID-19 Vaccine; Remdesivir; Antibiotics
MeSH Terms: conditions — Breast Feeding; COVID-19 | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The following samples may be collected:
  * Human Milk
  * Deciduous teeth from your breastfed children
  * Saliva Samples
  * Nostril Swabs
  * Stool Samples
  * Blood Samples (finger-prick)
  * Home Environmental Swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Main Study: The purpose of this project is to collect and store breast milk samples and health information about moms and their babies in a Human Milk Biorepository at UCSD. Through these studies, researchers hope to understand more about the benefits of breast milk, and how it prevents or treats child health problems.
- Sub-study 100: COVID-19 Exposure: The purpose of this substudy is to learn how exposures to COVID-19 and breastfeeding may affect the development of the child. Women who contact the UCSD Human Milk Biorepository will be screened for possible COVID-19 infection or exposure. Women will be eligible to enroll in the COVID-19 sub-study if they are confirmed positive, are presumptive positive, are symptomatic but not tested, or have confirmed exposure but are asymptomatic.
  Interventions: Biological: COVID-19 Exposure
- Sub-study 101: Antibiotic Exposure: The purpose of this substudy is to learn more about maternal use of antibiotics in women who do or do not breastfeed, and how this may influence infant and child health. Women who contact or are referred to the UCSD Human Milk Biorepository will be screened to participate in the Antibiotic Exposure sub-study. Women will be eligible to enroll in the Antibiotic Exposure sub-study if they are 18 years of age or older, have a singleton infant who is <3 months of age at the time of recruitment, and agree to all requirements of the study.
  Interventions: Drug: Antibiotic
- Sub-study 102: P50 MPRINT Admin Supplement: The purpose of this substudy is to review maternal medical exposure and how that may impact various components of human milk, the bacteria in the breastfed infant's gut, and the overall health and development of the breastfeeding child.

INTERVENTIONS:
Biological: COVID-19 Exposure — Have been or may have been exposed to COVID-19.
  Groups: Sub-study 100: COVID-19 Exposure
Drug: Antibiotic — Have or have not been prescribed one of several commonly used antibiotics including azithromycin, amoxicillin and clavulanic acid, amoxicillin, or nitrofurantoin.
  Groups: Sub-study 101: Antibiotic Exposure

SUMMARY:
The purpose of the UCSD Human Milk Biorepository is to establish and maintain a repository of breast milk samples that can be used to learn more about how breast milk influences infant and child health.

DETAILED DESCRIPTION:
Participants in this study will participate in the following:

1. Provide a milk sample:

   If participants agree, the investigators will ask participants to express 50ml (about 2 ounces) of milk. The investigators will take as much as participants wish to donate, or as little as one teaspoon.
2. Answer questions about participant's health:

   Future researchers may need to know if participants have any health problems, or about any treatments participants have had while breastfeeding. The investigators will ask participants for some contact information, health habits, and family's health history.
3. Fill out online questionnaires about participant's eating habits and mood:

   The investigators will ask the participant to answer an online questionnaire about how often participants eat certain foods.

   The investigators will also have the participant answer some questions about the participant's mood and how the participant has been feeling recently. The questionnaires can be completed on a tablet at the visit, or the investigators may send an email with a link to fill it out online. These questionnaires take about 30 minutes altogether.
4. The investigators will store the participant's sample and information in the Human Milk Biorepository:

   The investigators will keep the participant's milk and health information in the Human Milk Biorepository. There is no limit on the length of time we will keep the milk and information. The investigators will keep them as long as they are useful, unless the participant asks to remove them.
5. The investigators will let researchers use the stored materials for approved research studies:

   Researchers can apply to study the samples and information stored in the Human Milk Biorepository.
6. If the participant agrees, the investigators may contact the participant with information about other research studies.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 years old or older
* Breastfeeding
* Producing sufficient breast milk to donate an excess to the Biorepository

Exclusion Criteria:

* Women under 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any woman who is 18 or older, interested in participating, and is producing sufficient breast milk to donate an excess to the Biorepository will be invited to participate. We may enroll breastfeeding women who are pregnant or women who are pregnant and intend to breastfeed upon birth. We will not exclude any breastfeeding woman based on age (as long as above the legal age of consent), medical condition, or any other factor.
  Women will not be excluded based on exposures or lack thereof. We are currently enrolling women who have been or are exposed to:
  * Prescription Medications
    * SSRIs
    * Monoclonal Antibody Medications (mABS)
    * All other Rx medications
  * Women residing in Southern CA with a baby <6 months of age
  * Marijuana
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-03-27 (Actual); Primary Completion 2040-03 (Estimated); Study Completion 2040-03 (Estimated)

PRIMARY OUTCOMES:
Human Milk Repository | 1 year
  Establish a human milk repository at UCSD
Develop, maintain and manage the Repository | Through study completion, an average of 2 years
  Develop, maintain and manage the Repository as a resource for investigators to conduct research on the health characteristics and benefits of human breast milk.

SECONDARY OUTCOMES:
Sub-study 100: COVID-19 Exposure | Through study completion, an average of 2 years
  Develop, maintain and manage collection of other specimens for evidence of exposure to SARS-CoV-2, the virus responsible for COVID-19 disease.
Sub-study 101: Antibiotic Exposure | Through study completion, an average of 2 years
  Determine the pharmacokinetics of commonly used antibiotics (e.g., azithromycin, amoxicillin and clavulanic acid, amoxicillin or nitrofurantoin) in human milk samples.
Sub-study 102: P50 MPRINT Admin Supplement | Through study completion, an average of 2 years
  Expand enrollment in the UC San Diego human milk research biorepository to include 300 new participants who will provide milk samples paired with maternal and infant blood, stool, skin swabs, and maternal saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chambers, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Bertrand K, Kelly A, Chambers CD. The Prevalence of Nonserious Events in a Cohort of Breastfed Infants. Breastfeed Med. 2023 Jan;18(1):43-47. doi: 10.1089/bfm.2022.0245. Epub 2022 Nov 28. PMID 36454186